CLINICAL TRIAL: NCT06881238
Title: The Impact of Hepatitis B Virus Infection on the Clinical Course of Inflammatory Bowel Disease in Egyptian Patients
Brief Title: Impact of Hepatitis B Virus on Inflammatory Bowel Disease
Status: Recruiting | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Rania Mamdouh Elkafoury, Lecturer of Tropical Medicine, Tanta University
Other Study IDs: 36264PR979/12/24
Record Dates: First submitted 2025-03-04; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Inflammatory Bowel Disease (IBD); Hepatitis B Virus
Keywords: Hepatitis b virus; Inflammatory bowel disease course
MeSH Terms: conditions — Inflammatory Bowel Diseases; Hepatitis B

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- IBD patients with positive HBV infection.: 81 IBD patients with positive HBV infection.
  Interventions: Other: History of IBD course and outcome in HBV patients
- IBD Patients with negative HBV infection: 81 IBD Patients with negative HBV infection
  Interventions: Other: History of IBD course and outcome in HBV patients

INTERVENTIONS:
Other: History of IBD course and outcome in HBV patients — Full history taking including:
  * Personal history (name, age, sex, occupation, residence, and marital state).
  * Complaint.
  * Age at diagnosis of IBD.
  * Medication history.
  * History of hospital admissions and disease flares.
  * Disease extent, location, and behavior. (Montreal classification, Truelove-Witts severity index).
  * Surgical history (intestinal resection in CD patients and total proctocolectomy in UC patients).
  * Follow up duration and mortality.
  * Data of endoscopic examination
  * Data of laboratory investigations (complete blood picture, HBV serology, liver and kidney function tests, erythrocyte sedimentation rate (ESR), and C-reactive protein (CRP)).

SUMMARY:
The goal of this observational retrospective study is to assess the impact of hepatitis B virus (HBV) infection on the clinical course and outcomes of inflammatory bowel disease (IBD) in Egyptian patients.

Researchers will compare the IBD extent, location, severity, and behavior between IBD patients with and without HBV infection.

Participants will be subjected to history-taking (history of hospital admission and disease flare, surgical history, medication history, follow-up duration, and mortality), clinical examination, laboratory investigations, abdominal ultrasonography, and endoscopic examination.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients older than 18 years.
* Patients with IBD are diagnosed by clinical, radiological, endoscopic, and histological criteria.

Exclusion Criteria:

* Patients aged < 18 years
* Unwilling to participate in our study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: IBD patients attending the Tanta Tropical Medicine Department, Faculty of Medicine.
Sampling Method: Probability Sample
Enrollment: 162 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients with severe IBD measured by Truelove-Witts severity index | through study completion, an average of 6 month
  comparing IBD extent, location, and behavior using Montreal classification, Truelove-Witts severity index between patients with and without HBV infection
Hospital admission rates in IBD patients | through study completion, an average of 6 month
  comparing IBD hospital admission rates between patients with and without HBV infection
number of IBD patients undergoing surgical treatment | through study completion, an average of 6 month
  comparing surgical treatment rates (intestinal resection in CD patients and total proctocolectomy in UC patients) for IBD between patients with and without HBV infection

SECONDARY OUTCOMES:
Disease flares rates in IBD patients | through study completion, an average of 6 months
  comparing IBD disease flare rate between patients with and without HBV infection.
mortality rates in IBD patients | through study completion, an average of 6 months
  comparing IBD mortality rates between patients with and without HBV infection.

CONTACTS AND LOCATIONS:
Overall Officials: Nabila A Elgazzar, MD, Study Director — Tropical medicine and infectious diseases Department, Faculty of Medicine, Tanta University
Locations (1):
- Tanta University Hospitals, Tanta, Gharbyea, Egypt